CLINICAL TRIAL: NCT02413671
Title: Short-term Effects of Lupin Versus Whey Protein on Glucose and Insulin Responses to a Standardized Meal in a Randomized Controlled Trial
Brief Title: The Role of Whey and Lupin in Glycemic Control (Nutritional Pre-Study)
Acronym: NPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DLR German Aerospace Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NPS
Record Dates: First submitted 2015-03-24; First posted 2015-04-10 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Whole Body Glucose and Insulin Metabolism
MeSH Terms: interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lupin Protein (Other): Subjects received a test meal rich in carbohydrates and supplemented with lupin protein.
  Interventions: Dietary Supplement: Lupin Protein
- Whey Protein (Other): Subjects received a test meal rich in carbohydrates and supplemented with whey protein.
  Interventions: Dietary Supplement: Whey Protein
- Reference (Other): Subjects received a test meal rich in carbohydrates not supplemented with any protein.
  Interventions: Other: Reference

INTERVENTIONS:
Dietary Supplement: Lupin Protein — Subjects received a standardized test meal rich in carbohydrates and supplemented with lupin protein.
  Arms: Lupin Protein
Dietary Supplement: Whey Protein — Subjects received a standardized test meal rich in carbohydrates and supplemented with whey protein.
  Arms: Whey Protein
Other: Reference — Subjects received a standardized test meal rich in carbohydrates and not supplemented with any protein.
  Arms: Reference

SUMMARY:
The study compared the acute effects of the supplementation of a standardized meal with either lupin or whey protein or no protein on the whole-body glucose and insuline metabolism.

DETAILED DESCRIPTION:
The nutritional pre-study had the following key objectives:

Primary objective:

- Lupin protein lowers the postprandial blood glucose level equivalent to or to a greater extent than whey protein.

Secondary objective:

- Lupin protein has an equivalent or a stronger insulinotropic effect than whey protein.

ELIGIBILITY:
Inclusion Criteria:

* Female and male volunteers
* Age: between 20 and 45 years
* Body mass index (BMI): 20-28 kg/m²
* Fasting blood glucose within normal ranges (70-99 mg/dl; 29-42 mmol/mol Hb)
* Glycated hemoglobin HbA1c within normal ranges (4-6%)
* Agreement and signed informed consent before the study

Exclusion Criteria:

* Diabetes mellitus
* Increased bleeding tendency (hemophilia, regular use of anticoagulants)
* Allergy to nuts, legume or milk protein
* Drug, medication or alcohol abuse (frequent consumption of more than 20-30g alcohol/day)
* Intake of medication during the study
* Smoker
* Competitive athletes
* Extreme eating habits (vegan, special diets)
* Any other condition classed as unsuitable by the executive medical director

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Blood Glucose Metabolism by Blood Glucose and Serum Insulin (composite) | up to 180 minutes after the test meal was finished

CONTACTS AND LOCATIONS:
Overall Officials: Jörn Rittweger, Prof. Dr., Study Director — DLR German Aerospace Center; Ann-Charlotte Ewald, Principal Investigator — DLR German Aerospace Center; Kathrin Schopen, M.Sc., Principal Investigator — DLR German Aerospace Center; Petra Frings-Meuthen, Dr., Principal Investigator — DLR German Aerospace Center